CLINICAL TRIAL: NCT00274534
Title: A Comparison of the Effects of Tiotropium (18 Mcg) Inhalation Capsule q.d. and Salmeterol (50 Mcg) Inhalation Aerosol b.i.d. on Arterial Blood Gases in a Double-blind, Double-dummy, 4-week Crossover Study in Patients With Chronic Obstructive Pulmonary Disease (COPD).
Brief Title: A Comparison of the Effects of Tiotropium Inhalation qd and Salmeterol Inhalation Bid on Arterial Blood Gases.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 205.234
Record Dates: First submitted 2006-01-09; First posted 2006-01-11 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Salmeterol Xinafoate

INTERVENTIONS:
Drug: Tiotropium
Drug: Salmeterol

SUMMARY:
To evaluate changes in PaO2 following inhalation of Tiotropium by HandiHaler compared to Salmeterol MDI in patients with moderate to severe COPD.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2000-12; Study Completion 2003-07

PRIMARY OUTCOMES:
The change from baseline (Visit 2) in the PaO2 area under the curve (AUC) for the time period 0 to 105 minutes obtained through arterial blood gases (ABGs) at the end of each treatment period. | up to day 90

SECONDARY OUTCOMES:
Maximum decline in PaO2 from baseline | up to day 90
Maximum increase in alveolar-arterial oxygen gradient from baseline | up to day 90
Change from baseline (Visit 2) in FEV1 prior to insertion of catheter and 15 minutes post removal of catheter | up to day 90
Change from baseline (Visit 2) in FVC prior to insertion of catheter and 15 minutes post removal of catheter | up to day 90
Rescue medication use | up to day 90
COPD symptom score | up to day 90
Occurrence of adverse events | up to day 90
Pulse rate and sitting blood pressure in conjunction with spirometry | up to day 90

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim
Locations (2):
- United States (2):
  - Hines Veterans Administration Hospital, Hines, Illinois
  - Hunter Holmes McGuire Medical Center, Richmond, Virginia